CLINICAL TRIAL: NCT06929572
Title: Autologous Human Umbilical Cord Tissue Patch for Postnatal Closure of Open Neural Tube Defects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Stephen Fletcher, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-24-1194
Record Dates: First submitted 2025-03-26; First posted 2025-04-16 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Spina Bifida
Keywords: open neural tube defects; autologous umbilical cord patch; myelomeningocele; myeloschisis
MeSH Terms: conditions — Spinal Dysraphism; Meningomyelocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous umbilical cord patch (Experimental)
  Interventions: Procedure: Autologous umbilical cord patch

INTERVENTIONS:
Procedure: Autologous umbilical cord patch — Surgery will occur from birth to 24 hours of age. The autologous umbilical cord patch is harvested at time of delivery and immediately processed in a sterile setting in order to create a dural patch as a spinal cord cover to close the developmental defect within a few hours after birth.

SUMMARY:
The purpose of this study is to determine the impact of an autologous umbilical cord patch for dural closure on the repair of open neural tube defect. The outcomes will evaluate successful defect closure, creation of a more capacious spinal canal, and reduction in inflammatory tissue response versus historical controls.

ELIGIBILITY:
Inclusion Criteria:

* Neonates born with prenatal diagnosis of open neural tube defect (myelomeningocele or myeloschisis)
* Resident of the United States
* Provision of signed and dated informed consent form
* Stated willingness by legally authorized representative (LAR) to comply with all study procedures and availability for the duration of the study
* Maternal age 18 years and older
* Mother is English or Spanish Speaking

Exclusion Criteria:

* Sepsis or signs of infection of the neonate
* Febrile or other acute illness of the neonate at time of delivery
* Major congenital anomaly unrelated to spina bifida that may impact safety of neonate for surgery
* Evidence of intra-amniotic or maternal infection related to pregnancy at time of delivery
* Maternal use of steroid therapy during pregnancy or neonate use of steroid therapy,except for lung maturity indications
* Vaginal delivery
* Patch closure of dura is deemed unnecessary
* Umbilical cord abnormality
* Insufficient autologous cord tissue or patch
* Autologous umbilical cord patch that does not meet laboratory safety standards per standard operating procedure (SOP)
* Treatment with an investigational drug or other intervention that would influence morbidity or mortality

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants that have wound dehiscence | one-month post-op
Number of participants that have wound dehiscence | 1-year post-op
Number of participants that have Cerebrospinal fluid (CSF) leakage | one-month post-op
Number of participants that have CSF leakage | 1-year post-op.

SECONDARY OUTCOMES:
Number of participants that present with tethered cord syndrome | one-month post-op,12-months post-op, 30-months post-op, and 60-months post-op
Number of participants that had a change in level of neurological function as assessed by the American Spinal Injury Association Impairment Scale (ASIA) | baseline, one-month post-op,12-months post-op

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Fletcher, DO, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No